CLINICAL TRIAL: NCT07051395
Title: Correlation Between Coagulation Profiles And Injury Severity In Road Traffic Accidents Patients at Dera Ismail Khan
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHSW/Batch-Fall23/922
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Accident, Traffic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Road Traffic Accidents Patient — Coagulation Profiles And Injury Severity In Road Traffic Accidents Patients at Dera Ismail Khan

SUMMARY:
Trauma-induced coagulopathy (TIC), also known as acute traumatic coagulopathy (ATC), is a common condition in patients with severe trauma, particularly in road traffic accident (RTA) victims. Coagulopathy is often associated with high mortality rates and poor outcomes in trauma patients.

DETAILED DESCRIPTION:
The study explores the correlation between coagulation profiles and the severity of injuries in patients admitted to a tertiary care hospital following RTAs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe injuries (Injury Severity Score>15).
* All Patients will be admitted in Accident and Emergency Center after the accident.

Exclusion Criteria:

* Patients with Mild injury and score <15.
* Patients with pre-existing coagulation disorders (e.g., hemophilia).
* Patients on anticoagulant therapy prior to admission.
* Patients with incomplete medical records or insufficient blood samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To assess the correlation between coagulation profiles and injury severity in trauma patients, with a focus on the prevalence of trauma-induced coagulopathy (TIC) in road traffic accident (RTA) cases at a tertiary care hospital in Dera Ismail Khan.
  Methods: A cross-sectional observational study will be conducted in the Accident & Emergency (A&E) Department and Trauma Center of DHQ Hospital, Dera Ismail Khan. The study population includes patients aged 18 years and above, with moderate to severe injuries (Injury Severity Score ≥ 15),
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Self Admisnistred questioner | 12 Months
  A Self Admisnistred questioner is used to collect the data and details of the accident

CONTACTS AND LOCATIONS:
Locations (1):
- Mufti Mehmood Memorial Teaching Hospital, Dera Ismāīl Khān, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No